CLINICAL TRIAL: NCT03038893
Title: Point of Care Ultrasound For The Diagnosis Of Deep Venous Thrombosis And Its Effect On Length Of Hospital Stay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 54321516.0.0000.5327
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Deep Venous Thromboses; Deep Venous Thrombosis of Left Leg; Deep Venous Thrombosis of Right Leg; Deep Venous Thrombosis Proximal
Keywords: Ultrasonography; Point-of-care systems; Deep venous thrombosis; Hospitalization
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single Blind Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POCUS + EDUS (Experimental): Patients were first submitted to Point Of Care Ultrasound (POCUS) and then to Echo Doppler Ultrasound (EDUS) for the diagnosis of DVT.
  Interventions: Diagnostic Test: Point Of Care Ultrasound (PODUS)
- Echo Doppler Ultrasound (EDUS) (Active Comparator): Patients were submitted only to Echo Doppler Ultrasound (EDUS) for the diagnosis of DVT.
  Interventions: Diagnostic Test: Echo Doppler Ultrasound (EDUS)

INTERVENTIONS:
Diagnostic Test: Point Of Care Ultrasound (PODUS) — Patients were first submitted to Point Of Care Ultrasound (POCUS) and then to Echo Doppler Ultrasound (EDUS) for the diagnosis of DVT.
  Arms: POCUS + EDUS
Diagnostic Test: Echo Doppler Ultrasound (EDUS) — Patients were submitted only to Echo Doppler Ultrasound (EDUS) for the diagnosis of DVT.
  Arms: Echo Doppler Ultrasound (EDUS)

SUMMARY:
This is a Clinical Trial on the use of Point Of Care Ultrasound for the diagnosis of deep venous thrombosis (DVT) and its effect on length of hospital stay. 25 participants with suspicion of DVT according to Wells Criteria were randomized to one of two groups: Point of Care Ultrasound and Echo Doppler Ultrasound (POCUS + EDUS), and the control group was submitted only to the Echo Doppler Ultrasound (EDUS). The primary outcome was hospital stay.

DETAILED DESCRIPTION:
Because of high mortality associated with venous thrombosis (pulmonary embolism and deep venous thrombosis - DVT) the early recognition and therapeutics of its condition are crucial. Point of Care Ultrasound (POCUS) is a method with high sensibility to diagnose DVT and it is as accurate as Echo Doppler Ultrasound (EDUS), however the use of POCUS for diagnosis of DVT in the emergency care still presents resistance. This is a Clinical Trial on the use of POCUS for the diagnosis of DVT and its effect on length of hospital stay. 25 participants were randomized into two groups. The randomization was done through the random.org site in blocks of 4, a randomization list was with one researcher (blind) of the study. The experimental group was first submitted to POCUS in the Emergency Room, performed by a resident physician of Internal Medicine with training in POCUS, then after submitted to EDUS in the Radiology Service by a Radiologist. The control group was submitted only to EDUS in the Radiology Service. The 2-point compression technique was used, as described in previous studies, using the portable ultrasound device (M-turbo Sonosite) with a high frequency linear transducer (5-10 MHZ). The sites used in the evaluation were the popliteal site comprising the popliteal vein and trifurcation of the popliteal vein and the femoral point in which comprises the sapheno-femoral junction, the common femoral vein and the superficial femoral vein, all evaluated in the transverse plane. The result was considered positive for DVT when the vessel evaluated showed no compressibility and / or presented echogenic material in the lumen of the vein. After the randomization, the patients were followed for a period of 30 days, being evaluated in three moments: initial evaluation, at 7 and 30 days of the initial evaluation. Whenever possible, each evaluation was in person. In the initial evaluation, the participant's demographics, date and time of arrival at the Emergency Service, previous illnesses, Wells criteria score and reason for the initial care were collected. Participants randomized to the POCUS + EDUS group had recorded date and time of ultrasound at the bedside and, if there was confirmation of DVT, these data were collected by the resident physician, blinded for the Echo Doppler Ultrasound results. EDUS data, such as date and time of the examination request, date and time of the release of the exam report, confirmation of DVT, date and time of discharge were collected by another researcher, blinded to the participant's group and to the POCUS's results. After 7 and 30 days the outcomes were recorded: time for a first diagnostic information, time to therapeutic decision making / prescription, length of hospital stay, death, pulmonary thromboembolism, bleeding or other complication, re-hospitalization, evolution to DVT in cases that were initially negative.

ELIGIBILITY:
Inclusion Criteria:

* Low, moderate or high suspicion of DVT by Wells Criteria.
* Patients with Echo-Doppler Ultrasonography already requested in the hospital system.

Exclusion Criteria:

* Myocardial Infarction, Stroke or Cardiac Surgery within 3 months prior to hospital admission;
* Renal Chronic Disease (Clinical Stages IV and V);
* Congestive Heart Failure (NYHA IV);
* Pregnancy;
* Previous episode of DVT in the same leg that of the current DVT suspicion;
* Patients already in treatment for DVT or taking anticoagulants for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Up to 30 days
  Length of hospital stay

SECONDARY OUTCOMES:
Time to first diagnostic information | Up to 30 days
  Time to first diagnostic information
Time to therapeutic decision making / prescription | Up to 30 days
  Time to therapeutic decision making / prescription

CONTACTS AND LOCATIONS:
Overall Officials: Ana Claudia Tonelli, Principal Investigator — Hospital de Clinicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided